CLINICAL TRIAL: NCT05702866
Title: Apport de l'évaluation de l'ischémie de Membre supérieur Par oxymétrie transcutanée Dans la caractérisation de la Compression Vasculaire Chez Les Patients Suspects de Syndrome du défilé Thoraco-brachial
Brief Title: Vascular Compression Assessment Using Transcutaneous Oxymetry in Patients Suspected of Having Thoracic Outlet Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-161
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Thoracic Outlet Syndrome
Keywords: transcutaneous oximetry; thoracic outlet syndrome; arteriography; vascular compression
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Suspected of Having Thoracic Outlet Syndrome: Patients who came for the diagnosis of TOS
  Interventions: Diagnostic Test: Transcutaneous oximetry

INTERVENTIONS:
Diagnostic Test: Transcutaneous oximetry — Comparison of the TcpO2 values recorded during dynamic maneuver with the estimated rate of compression of the subclavian and axillary vessels determined on dynamic angiography.

SUMMARY:
Thoracic outlet syndrome (TOS) is characterized by nervous, venous or arterial symptoms resulting from a compression of the thoracic bundle in the thoracic outlet. The diagnostic approach of TOS is still controversial. The investigating team is interested in arterial TOS and have already been able to demonstrate the presence of arm ischemia during dynamic maneuvers using transcutaneous oximetry (TcpO2). The correlation between the measurement of TcpO2 during dynamic maneuvers and the vascular compression type (arterial, venous or both) will be evaluated. The evaluation the correlation between TcpO2 and degree of arterial compression observed in dynamic arteriography (considered as a gold standard examination) will be calculated too. The use of TcpO2 could be developed in the diagnosis assessment of TOS.

ELIGIBILITY:
Inclusion Criteria:

* patient suspected of having a thoracic outlet syndrome
* patient having carried out additional examinations as part of the diagnostic assessment : venous and arterial Doppler or dynamic arteriography and venography
* patient having carried out a dynamic TcpO2 recording

Exclusion Criteria:

* patient under 18 year old
* non french speaker
* patient who expressed his/her refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting to the vascular medicine department with suspected thoracic outlet syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
DROPmin according on the type of compression | thirty minutes
  Variation in upper limb ischemia is estimated by TcpO2 measurement and calculating of the DROPmin (TcpO2 variation regarding a reference) depending on the type of damage (arterial, venous, or both arterial and venous).
  DROP is Decrease Rest of Oxygen Pressure

SECONDARY OUTCOMES:
DROPmin according on the degree of arterial stenosis | thirty minutes
  To assess the correlation between the severity of upper limb ischemia by TcpO2 measurement and the degree of arterial stenosis observed in diagnostic arteriography.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No